CLINICAL TRIAL: NCT05194930
Title: A Novel Acceptance-based Treatment for Insomnia in Veterans With Post-Traumatic Stress Disorder
Brief Title: Treatments for Insomnia in Veterans With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 20-283
Record Dates: First submitted 2022-01-05; First posted 2022-01-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; PTSD
Keywords: Insomnia disorder; Chronic Post-Traumatic Stress Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded from group assignment and the treatment content. Participants will be blinded to the content of the treatment arm to which they are not assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The ABC of Insomnia (Acceptance and the Behavioral Changes to (Experimental): This is the new treatment arm that is being compared to CBT-I, standard treatment for insomnia.
  Interventions: Behavioral: The ABC of Insomnia (Acceptance and the Behavioral Changes to treat Insomnia)
- Cognitive-Behavioral Therapy for Insomnia (Active Comparator): This is the standard treatment for insomnia that is being compared to the new treatment (ABCI).
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: The ABC of Insomnia (Acceptance and the Behavioral Changes to treat Insomnia) — 5 individual sessions incorporating behavioral treatment components plus acceptance and commitment therapy (ACT) provided by a trained instructor.
  Other Names: ABC-I
  Arms: The ABC of Insomnia (Acceptance and the Behavioral Changes to
Behavioral: Cognitive-Behavioral Therapy for Insomnia — 5 individual sessions incorporating behavioral and cognitive therapy components with a trained instructor.
  Other Names: CBT-I
  Arms: Cognitive-Behavioral Therapy for Insomnia

SUMMARY:
This randomized trial will compare a novel treatment, Acceptance of the Behavioral Changes to Treat Insomnia (ABC-I) to Cognitive Behavioral Therapy for Insomnia (CBT-I) among Veterans with comorbid Post-Traumatic Stress Disorder (PTSD) and insomnia disorder. ABC-I combines the behavioral components of CBT-I with components of another behavioral therapy (Acceptance and Commitment Therapy) and has been shown to improve treatment adherence.

The study objectives are: 1) to evaluate the benefits of ABC-I in reducing post-traumatic stress disorder (PTSD) symptoms among Veterans with comorbid PTSD and insomnia disorder compared to CBT-I, and 2) to evaluate the effectiveness of ABC-I in improving insomnia symptoms and sleep quality among Veterans with comorbid PTSD and insomnia disorder as compared to CBT-I.

Veterans with insomnia and comorbid PTSD who receive care at Sepulveda and West Los Angeles facilities will be recruited for the study. Those who pass an initial eligibility screen will be enrolled and written informed consent will be obtained. A baseline assessment will be completed that includes measures of sleep, PTSD, and quality of life. Veterans who meet all eligibility criteria will be randomly assigned to the ABC-I (n=100) or CBT-I (n=100) treatment. Both treatments will be provided in 5 one-on-one sessions by a trained instructor who is supervised by a behavioral sleep medicine specialist. All randomized participants (n=200) will have 3 follow-up assessments (post-treatment, 3-months, and 6-months after randomization). The follow-up assessments will collect information on PTSD symptoms, insomnia symptoms and sleep quality.

DETAILED DESCRIPTION:
Poor sleep is a nearly universal experience after trauma and in the context of PTSD non-pharmacological therapies are considered first-line treatments, yet VA/DoD clinical practice guidelines acknowledged the paucity of available evidence on the treatment of insomnia disorder in the context of PTSD. There is evidence of sleep-related benefits with CBT-I for individuals with insomnia and psychiatric comorbidities, but challenges remain. Insomnia treatments studied among Veterans with PTSD have typically been combined treatments to address both conditions. While promising, these treatments are difficult to implement because of their length and complexity. Furthermore, studies generally have not compared novel sleep-focused treatments to CBT-I (i.e., standard care for insomnia), making it difficult to support a change in the allocation of clinical resources to train providers in new sleep-focused interventions.

This randomized trial will compare a novel treatment, Acceptance of the Behavioral Changes to Treat Insomnia (ABC-I) to Cognitive Behavioral Therapy for Insomnia (CBT-I) among Veterans with comorbid Post-Traumatic Stress Disorder (PTSD) and insomnia disorder. ABC-I combines the behavioral components of CBT-I with components of another behavioral therapy (Acceptance and Commitment Therapy) and has been shown to improve treatment adherence.

The study objectives are: 1) to evaluate the benefits of ABC-I in reducing PTSD symptoms among Veterans with comorbid PTSD and insomnia disorder compared to CBT-I, and 2) to evaluate the effectiveness of ABC-I in improving insomnia symptoms and sleep quality among Veterans with comorbid PTSD and insomnia disorder as compared to CBT-I.

Veterans with insomnia and comorbid PTSD who receive care at Sepulveda and West Los Angeles facilities will be recruited for the study. Those who pass an initial eligibility screen will be enrolled and written informed consent will be obtained. A baseline assessment will be completed that includes measures of sleep, PTSD, and quality of life. Veterans who meet all eligibility criteria will be randomly assigned to the ABC-I (n=100) or CBT-I (n=100) treatment. Both treatments will be provided in 5 one-on-one sessions by a trained instructor who is supervised by a behavioral sleep medicine specialist. All randomized participants (n=200) will have 3 follow-up assessments (post-treatment, 3-months, and 6-months after randomization). The follow-up assessments will collect information on PTSD symptoms, insomnia symptoms and sleep quality. The analytic plan will simultaneously address superiority of ABC-I over CBT-I for improving PTSD symptoms and non-inferiority of ABC-I compared to CBT-I for improving insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling Veterans aged 18 years and older,
* received care from VAGLAHS in the prior year,
* live within a 50-mile radius of the research offices at the VA Sepulveda Ambulatory Care Center,
* have symptoms of PTSD,
* have symptoms of insomnia.

Exclusion Criteria:

* current pregnancy or has a child less than 6 months of age (men and women),
* active substance users or in recovery with less than 90 days of sobriety,
* too ill to engage in the study procedures,
* unable to self-consent to participate,
* unstable housing (since we may not be able to retrieve costly and difficult to replace monitoring equipment),
* severe, untreated sleep disordered breathing (AHI>15 with excessive daytime sleepiness, or AHI>30),
* restless legs syndrome that accounts for the sleep disturbances reported,
* a circadian rhythm sleep disorder that accounts for the sleep disturbances reported (including shift work sleep disorder),
* unstable medical or psychiatric disorders (which is a contraindication for behavioral treatment of insomnia);
* remission of insomnia symptoms prior to randomization;
* current participation in prolonged exposure therapy for PTSD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Check List for DSM-5 (PCL-5) | 6-months follow-up
  The PCL-5 total score will be the main outcome measure for PTSD symptom severity. The PCL-5 is a standardized assessment for PTSD, based on DSM-5. The 20-item scale assesses the presence and severity PTSD symptoms on a 0-4 Likert scale, with a total symptom severity score range from 0-80. A score greater than or equal to 33 is indicative of probable PTSD.
Insomnia Severity Index (ISI) | 6-months follow-up
  Mean score on Insomnia Severity Index (ISI). This 7-item scale measures self-reported severity of insomnia symptoms.
  Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Pittsburgh Sleep Quality Index (PSQI) | 6-months follow-up
  Mean PSQI score will be used as a measure of sleep quality. Scores range from 0 to 21. Higher scores indicate worse sleep quality.
Sleep efficiency from 7-day sleep diary | 6-months follow-up
  Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of self-reported sleep diary.
  Scores range from 0 to 100 percent. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Martin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson GC, Kelly MR, Mitchell M, Josephson KR, McGowan SK, Culver NC, Kay M, Alessi CA, Fung CH, Washington DL, Hamilton A, Yano EM, Martin JL. Benefits of Cognitive Behavioral Therapy for Insomnia for Women Veterans with and without Probable Post-Traumatic Stress Disorder. Womens Health Issues. 2022 Mar-Apr;32(2):194-202. doi: 10.1016/j.whi.2021.10.007. Epub 2021 Nov 21. PMID 34815139
- [Background] Martin JL, Carlson GC, Kelly MR, Song Y, Mitchell MN, Josephson KR, McGowan SK, Culver NC, Kay MA, Erickson AJ, Saldana KS, May KJ, Fiorentino L, Alessi CA, Washington DL, Yano EM. Novel treatment based on acceptance and commitment therapy versus cognitive behavioral therapy for insomnia: A randomized comparative effectiveness trial in women veterans. J Consult Clin Psychol. 2023 Nov;91(11):626-639. doi: 10.1037/ccp0000836. Epub 2023 Aug 3. PMID 37535521